CLINICAL TRIAL: NCT07021261
Title: A Multicenter, Open-Label, Randomized, Phase III Study Comparing UTD2 Combined With Capecitabine to Capecitabine Monotherapy as Adjuvant Therapy for Triple-Negative Breast Cancer Patients Who Did Not Achieve Pathological Complete Response
Brief Title: Comparing UTD2 Combined With Capecitabine to Capecitabine as Adjuvant Therapy for Non-pCR TNBC Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of the Department of Breast Surgery, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG02-T2401
Record Dates: First submitted 2025-05-18; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; TNBC
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Utidelone plus capecitabine (Experimental): UTD2 50 mg/m²/day orally on Days 1-5, repeated every 21 days for 2 years; Capecitabine 1000 mg/m² twice daily on Days 1-14, repeated every 21 days for 8 cycles.
  Interventions: Drug: Utidelone plus capecitabine
- Capecitabine (Active Comparator): Capecitabine 1000 mg/m² twice daily on Days 1-14, repeated every 21 days for 8 cycles.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Utidelone plus capecitabine — UTD2 50 mg/m²/day orally on Days 1-5, repeated every 21 days for 2 years; Capecitabine 1000 mg/m² twice daily on Days 1-14, repeated every 21 days for 8 cycles.
  Other Names: UTD2 plus capecitabine
  Arms: Utidelone plus capecitabine
Drug: Capecitabine — Capecitabine 1000 mg/m² twice daily on Days 1-14, repeated every 21 days for 8 cycles.
  Arms: Capecitabine

SUMMARY:
Evaluate the IDFS rate, overall survival (OS) rate, and safety profile of UTD2 combined with capecitabine versus capecitabine monotherapy as adjuvant therapy for triple-negative early breast cancer patients who did not achieve pathological complete response (pCR) after neoadjuvant therapy.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label phase III clinical study that aims to evaluate the efficacy and safety of the combination therapy involving the use of oral UTD2 capsule in conjunction with capecitabine, as compared to the efficacy and safety of capecitabine monotherapy. The study is specifically focused on patients diagnosed with triple-negative early breast cancer who, after undergoing neoadjuvant therapy, did not achieve a pathological complete response (pCR). The primary objective of this research is to assess whether the addition of UTD2 to capecitabine can provide a more effective adjuvant treatment option for this particular group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent and Compliance The patient has fully understood this study and voluntarily signed the informed consent form, demonstrating the ability and willingness to comply with the study protocol-defined visits, treatment plans, laboratory tests, and other study procedures.
2. Age and Gender Female patients aged 18 to 70 years old (inclusive) on the day of signing the informed consent.
3. Prior Neoadjuvant Chemotherapy without pCR Received prior neoadjuvant chemotherapy containing anthracycline or taxane agents without achieving pathological complete response (pCR).

   Neoadjuvant chemotherapy requirement: At least 4 completed cycles. Non-pCR definition: Residual invasive carcinoma confirmed by pathology after primary tumor resection.
4. Surgical Resection Underwent complete surgical resection (R0) with pathologically confirmed negative margins.
5. Triple-Negative Breast Cancer Confirmation

   Post-resection tumor tissue confirmed as ER-negative, PR-negative, and HER2-negative breast cancer by immunohistochemistry (IHC):

   ER-negative: <1% expression by IHC. PR-negative: <1% expression by IHC. HER2-negative: IHC score of 0 or 1+, or 2+ with negative in situ hybridization (ISH) results.
6. Postoperative Treatment No prior systemic anticancer therapy (excluding radiotherapy) after breast cancer surgery.
7. Performance Status ECOG performance status of 0 to 1.
8. Hematological Criteria (within 1 week prior to enrollment)

   Blood tests meet the following criteria (CTCAE v5.0 ≤ Grade 1, based on institutional laboratory standards):

   White blood cell (WBC) count ≥ 3.0 × 10^9/L. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L. Platelet (PLT) count ≥ 100 × 10^9/L. Hemoglobin ≥ 9.0 g/dL. No administration of recombinant human granulocyte colony-stimulating factor (rhG-CSF), blood products, or erythropoietin (EPO) within 14 days prior to enrollment.
9. Biochemical Criteria (within 1 week prior to enrollment)

Normal blood biochemistry (CTCAE v5.0 ≤ Grade 1, based on institutional laboratory standards):

Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN). Alanine aminotransferase (ALT) ≤ 1.5 × ULN. Aspartate aminotransferase (AST) ≤ 1.5 × ULN. Alkaline phosphatase (ALP) ≤ 2.5 × ULN. Creatinine clearance (Ccr) ≥ 50 mL/min. Contraception Requirements Fertile patients must agree to use highly effective contraception (hormonal, barrier methods, or abstinence) with their partners during the trial and for at least 6 months after the last dose. Premenopausal female patients must have a negative blood or urine pregnancy test before enrollment.

Exclusion Criteria:

1. Stage IV metastatic breast cancer.
2. Bilateral breast cancer.
3. History of other malignancies within the past 5 years, except for cured basal cell carcinoma of the skin, cervical carcinoma in situ, or papillary thyroid carcinoma.
4. Radiotherapy within 2 weeks prior to the first dose of the study drug.
5. Surgery within 2 weeks prior to the first dose of the study drug.
6. Prior treatment with utidelone or capecitabine, known hypersensitivity to utidelone, capecitabine, or fluoropyrimidines, or confirmed dihydropyrimidine dehydrogenase (DPD) deficiency.
7. Prior adverse reactions to anticancer therapy have not recovered to CTCAE v5.0 Grade ≤1 (excluding toxicities deemed non-risky by the investigator, such as alopecia).
8. Gastrointestinal disorders (e.g., esophageal obstruction, pyloric obstruction, intestinal obstruction), post-gastrointestinal resection, or other factors causing dysphagia that may interfere with oral drug absorption.
9. Severe comorbidities, including significant cardiac/cerebrovascular disease, uncontrolled diabetes/hypertension, active infections, or active peptic ulcer.
10. Active hepatitis B virus (HBV) infection.
11. History of immunodeficiency (e.g., HIV-positive status, congenital/acquired immunodeficiency disorders) or organ transplantation.
12. Psychiatric disorders or poor compliance.
13. Pregnancy (positive pregnancy test) or lactation.
14. Concurrent participation in another interventional clinical study or receiving other investigational therapies.
15. Concomitant use of potent CYP3A4 inhibitors/inducers or QT-prolonging drugs within 14 days prior to the first dose or during the study.
16. Other conditions deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2030-06-16 (Estimated); Study Completion 2032-06-16 (Estimated)

PRIMARY OUTCOMES:
3-year invasive disease-free survival(IDFS) | 36 months
  defined as occurrence of any of the following: ipsilateral invasive breast cancer recurrence, regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer, or second non-breast invasive cancer.In-situ events are not included.

SECONDARY OUTCOMES:
invasive disease-free survival(IDFS) | 60 months
  defined as occurrence of any of the following: ipsilateral invasive breast cancer recurrence, regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer, or second non-breast invasive cancer.In-situ events are not included.
overall survival (OS) | 36 months
  the time from treatment to death, regardless of disease recurrence
overall survival (OS) | 60 months
  the time from treatment to death, regardless of disease recurrence
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 months
  Collect all participants' adverse event data and classify and assess them according to the CTCAE v4.0 criteria. This includes documenting the type of adverse event, severity (Grade 1-5), duration, and whether it is related to the study treatment. Data collection can be conducted through electronic health records, patient reports, or investigator reports, among other methods.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT07021261/Prot_SAP_000.pdf